CLINICAL TRIAL: NCT06534788
Title: Effects of Reciprocal Inhibition Versus Post Facilitation Muscle Energy Technique Along With Conventional Physical Therapy in Patients With Piriformis Syndrome: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/21
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: This will be a single blinded study because the treatment of both study group and control group will be done by the researcher and only the participants will be kept blinded about the allocation of participants to either the active comparator group or experimantal group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RI-MET group (Experimental): RI-MET group A will receive 3-5 repetitions of reciprocal inhibition to the shortened piriformis muscle in supine and prone positions i.e. 30-50% isometric contraction of the muscle opposite to the muscle to be stretched for 7-10 seconds, followed by inhalation, exhalation and rest period of 5 seconds and then a stretch (through the new barrier with patients' assistance) of 10-60 seconds hold.both groups will receive conventional physical therapy which they will be taught as a home plan. Following exercises are guided to the patient as home plan.
  * Resisted abduction with Thera/resistance band
  * Resisted bridging with Thera/resistance band
  * Resisted clam exercise with Thera/resistance band
  Interventions: Other: Reciprocal Inhibition MET; Other: Conventional physical therapy
- PFS-MET group (Experimental): PFS-MET group will receive 3-5 repetitions of post-facilitation stretch to the shortened piriformis muscle in supine and prone positions i.e. 20% maximal isometric contraction of the muscle to be stretched for 6-10 seconds, followed by a rapid stretch (through the new barrier) of 15 seconds hold.
  After stretch, the muscle is allowed to relax in the midrange for up to 30 seconds.Both groups will receive conventional physical therapy which they will be taught as a home plan. Following exercises are guided to the patient as home plan.
  * Resisted abduction with Thera/resistance band
  * Resisted bridging with Thera/resistance band
  * Resisted clam exercise with Thera/resistance band
  Interventions: Other: Post-facilitation MET; Other: Conventional physical therapy

INTERVENTIONS:
Other: Reciprocal Inhibition MET — Reciprocal Inhibition MET will be applied to the shortened piriformis muscle in supine and prone positions with participants using 30-50% of their maximum voluntary isometric contraction. It will include 30-50% isometric contraction of the muscle opposite to the muscle to be stretched for 7-10 seconds, followed by inhalation, exhalation and rest period of 5 seconds and then a stretch (through the new barrier with patients' assistance) of 10-60 seconds hold. RI-MET group will receive 3-5 repetitions.
  Arms: RI-MET group
Other: Post-facilitation MET — Post-facilitation stretch technique for shortened piriformis muscle in supine and prone positions will be applied with participants using 20% of their maximum voluntary isometric contraction. It will include 20% maximal isometric contraction of the muscle to be stretched for 6-10 seconds, followed by a rapid stretch (through the new barrier) of 15 seconds hold. After stretch, the muscle is allowed to relax in the midrange for up to 30 seconds. PFS-MET group will receive 3-5 repetitions.
  Arms: PFS-MET group
Other: Conventional physical therapy — TENS and hot pack application to provide heating effect over the painful area (10 minutes) Both groups will receive conventional physical therapy which they will be taught as a home plan. Following exercises are guided to the patient as home plan.
  * Resisted abduction with Thera/resistance band
  * Resisted bridging with Thera/resistance band
  * Resisted clam exercise with Thera/resistance band

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to compare the effects of reciprocal inhibition versus post facilitation muscle energy technique along with conventional physical therapy in patients with piriformis syndrome in terms of pain, range of motion at hip joint and functional disability.

DETAILED DESCRIPTION:
This study aims to compare the effects of reciprocal inhibition with post facilitation muscle energy technique along with conventional physical therapy in terms of pain, functional disability and range of motion at hip joint in patients with piriformis syndrome to find the best suitable and effective treatment for it based on the outcomes.

Males and females between the age of 20-50 years, having buttock pain of ≥ 3 on NPRS since 3 months or more and a score of ≥ 8 on a 12-point clinical scoring system as well as any two of the positive screening tests will be recruited in this study as patients of piriformis syndrome.

These subjects will be selected via non-probability purposive sampling technique, followed by randomization into two groups using blocked randomization method.

A total of 6 treatment sessions will be given to each participant over the duration of 2 weeks with a total of 3 follow-ups after every 2 sessions.

TENS and hot pack followed by reciprocal inhibition technique will be given to the experimental group A, while the active comparator group B will be given TENS and hot pack followed by post-facilitation muscle energy technique.

Both the groups will be guided about the strengthening exercises given as a home plan.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years
* Both Genders
* Chronic pain in buttock and hip area (≥ 3 on NPRS) lasting more than 3 months.
* Shortened piriformis muscle (Internal rotation less than 30°) on muscle length assessment.
* A score of ≥ 8 on a 12-point clinical scoring system.
* At least two positive screening tests.

Exclusion Criteria:

* Active infection
* Lower lumbar radiculopathy
* Sacroiliac joint dysfunction
* Malignancies
* History of trauma
* Hip Arthroplasty
* Rheumatoid/ Osteoarthritis
* Any neurological dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 2 weeks
  The pre and post pain intensity will be measured using Numeric Pain Rating Scale (NPRS) comprising of 11 points from 0 - 10 where 0 indicates "no pain" while 10 is "maximally felt pain".
Hip range of motion | 2 weeks
  Goniometer will be used to measure the pre and post treatment ranges of internal rotation, external rotation, abduction and adduction at hip joint in supine and sitting positions.
Functional Disability | 2 weeks
  Lower Extremity Functional Scale comprising of 20 questions regarding lower extremity function will be used. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan